CLINICAL TRIAL: NCT05339633
Title: An Open Label Phase 1 Study in Healthy Adult Female Subjects to Determine the Mass Balance Recovery, Absorption, Metabolism, and Excretion of [14C]-D-0502 Following Single Oral Dose Administration
Brief Title: Study in Healthy Adult Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D0502-103
Record Dates: First submitted 2022-03-25; First posted 2022-04-21 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Mass Balance Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Dose (Other): All study subjects will receive a a single oral dose of radiolabeled microtracer of D-0502 following an overnight fast
  Interventions: Drug: [14C]-D-0502

INTERVENTIONS:
Drug: [14C]-D-0502 — Drug: [14C]-D-0502 and D-0502

SUMMARY:
An Open Label Phase 1 Study in Healthy Adult Female Subjects to Determine the Mass Balance Recovery, Absorption, Metabolism, and Excretion of [14C] D-0502 Following Single Oral Dose Administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female volunteers not of child-bearing potential between the ages of 18 and 65. Other inclusion criteria will be reviewed by the Principal Investigator.

Exclusion Criteria:

* History or presence of any condition or prior surgery that, in the opinion of the Investigator, poses a significant risk to subject safety and/or achievement of study objectives
* Clinically significant abnormal medical history, or any abnormal findings on physical examination, vital signs, ECG, or laboratory tests
* Other exclusion criteria will be reviewed by the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Radiolabel recovery | 14 days
  To assess the mass balance (i.e., cumulative excretion in urine and feces) of D 0502 and the percentages of radiolabel recovered in urine and feces following administration of a single oral dose of D-0502/5 microcuries (µCi) [14C] D-0502 in healthy, adult female subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Site Location, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No